CLINICAL TRIAL: NCT05297006
Title: Regulation and Mechanism of New Compound Functional Ingredients on Intestinal Microecology and Immune Function in Infants
Brief Title: Regulation and Mechanism of New Compound Functional Ingredients in Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S170003
Record Dates: First submitted 2020-12-06; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Sialic Acid; Oligosaccharide
Keywords: Infant; Human milk; Growth and development; immune level
MeSH Terms: interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — breast milk, infants' blood, infants' faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breastfeeding group: The mother can breastfeed exclusively until the infants is at least 4 months old, after which complementary foods are added scientifically according to the baby's condition.
- Formula group containing new compound functional ingredients: Only use formula milk powder containing oligosaccharides, sialic acid and other ingredients feed the infants for at least 4 months, and then complementary food is added scientifically according to the infant's condition.
  Interventions: Dietary Supplement: The infants who drank milk powder were given a dietary intervention four months before
- Formula group without new compound functional ingredients: Only use formula milk powder without oligosaccharides, sialic acid and other ingredients feed the infants for at least 4 months, and then complementary food is added scientifically according to the infant's condition.
  Interventions: Dietary Supplement: The infants who drank milk powder were given a dietary intervention four months before

INTERVENTIONS:
Dietary Supplement: The infants who drank milk powder were given a dietary intervention four months before — The infants who eat milk powder were randomly divided into two groups: group containing new compound functional ingredients and group without new compound functional ingredients
  Groups: Formula group containing new compound functional ingredients; Formula group without new compound functional ingredients

SUMMARY:
A prospective, multicentre, randomized, double-blind, parallel control study was conducted to analyze the changes in growth, intestinal flora, and immune function of infants with different feeding patterns from postnatal to 1 year of age.

DETAILED DESCRIPTION:
Breast milk is the most beneficial and safe natural food for the growth and development of infants, but some mothers cannot complete breast feeding.For infants who cannot be breastfed, how to improve the composition of formula milk powder and improve the growth and development of infants is an important issue to be solved urgently in this field.It has been found that new compound functional ingredients oligosaccharides and sialic acid may be beneficial to the healthy growth and development of infants and young children, but the specific mechanism and significance are still unclear due to the lack of systematic research.Known as the "second Brain", the gut is connected to the Brain via the brain-gut-axis.Intestinal microecological status can significantly affect the development of infant nervous system and immune system, and then affect the occurrence of related diseases in adulthood.Oligosaccharides and sialic acid may affect the structure of intestinal microecology, protect the immune function of infants and promote the healthy development of infants.This project is based on the previous studies, using multicenter, prospective, randomized, double-blind, parallel-group trial, discussion of oligosaccharides and sialic acid in infants and young children the intestinal micro ecology and the regulation of immune function and the role mechanism, revealing the oligosaccharides and sialic acid in infants and young children the role of immediate and long-term growth, and the significance of these new type of composite function is added to the dairy ingredients, to research and development more accord with our country new dairy products provide theoretical basis for the healthy growth of infants and young children.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants;
2. Full-term (gestational age ≥37 weeks);
3. Birth weight 2500-4500g;
4. Mothers have no history of diabetes, hypertension, heart disease, and other diseases during pregnancy;
5. The guardian signed informed consent and voluntarily enrolled into the group and promised to complete systematic follow-up.

Exclusion Criteria:

1. Hospitalization with cognitive impairment or deformity ≥2 days
2. History of birth asphyxia (Apgar score < 3)
3. Severe allergy to milk and serious medical conditions such as intracranial hemorrhage, chronic diarrhea, necrotizing colitis, or acute infection
4. The guardian refused to enroll or could not complete the system follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Breastfeeding group The mother can breastfeed exclusively until the infants is at least 4 months old, after which complementary foods are added scientifically according to the baby's condition.
  Formula group containing new compound functional ingredients Only use formula milk powder containing oligosaccharides, sialic acid and other ingredients feed the infants for at least 4 months, and then complementary food is added scientifically according to the infant's condition.
  Formula group containing new compound functional ingredients Only use formula milk powder containing oligosaccharides, sialic acid and other ingredients feed the infants for at least 4 months, and then complementary food is added scientifically according to the infant's condition.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth and development indexes | 12 months
  Baby body length, weight, head circumference gain
Growth and development indexes | 12 months
  Baby body weight gain
Growth and development indexes | 12 months
  Baby body head circumference gain
Neurodevelopmental level | 4 months
  The Peabody scale was used to assess the level of neural development of infants at 4 months and 6 months
Neurodevelopmental level | 6 months
  The Peabody scale was used to assess the level of neural development of infants at 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided